CLINICAL TRIAL: NCT01413490
Title: A Clinical Study to Evaluate the Biological Effects of Administering Rimantadine in Patients With Hepatitis C Virus (HCV) Infection Alongside Standard Combination Therapy With Pegylated Interferon and Ribavirin
Brief Title: Hepatitis C Rimantadine and Antiviral Combination Therapy
Acronym: HepRiACT
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Lynsey Corless, doctor, The Leeds Teaching Hospitals NHS Trust
Other Study IDs: 2011-002781-21
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C
Keywords: hepatitis C virus; Interferon; rimantadine; liver
MeSH Terms: conditions — Hepatitis C | interventions — Rimantadine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples of patients undegoing standard combination therpay for hepatits c virus infection
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rimantadine — 12 weeks of rimantadine therapy in addition to standard combination therapy with interferon and ribavirin

SUMMARY:
Hepatitis C virus is one of the leading causes of liver failure and liver cancer worldwide. Current treatment of hepatitis C infection is only successful in about half of those who are eligible. The current treatment aims to boost the host immune system but does not directly act on the virus. Many drugs are in various stages of development that target the virus directly - their specific mode of action is confirmed by showing the virus is forced to adapt in the presence of the drug. As with many viruses, treating with only one specific drug would quickly lead to the virus adapting and becoming resistant. We therefore need to find new combinations of directly acting drugs. Rimantadine has already been shown in the laboratory to target hepatitis C directly. We have designed this study to see if it happens in real life as well. If so, we could use rimantadine to help fight hepatitis c more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of HCV infection, genotype 1 or genotype 3
* Be eligible for standard combination therapy with pegylated IFN and ribavirin
* Be at least 18 but no more than 65 years of age
* Have signed an informed consent indicating that the patient is aware of the infectious nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts
* Be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests
* Have no contraindications to receiving rimantadine therapy
* Have blood results within defined acceptable haematological and biochemical parameters (haemoglobin >10 g/dl, platelet count >150 x 109/L, bilirubin <25 umol/L, albumin >35 g/L, creatinine <150 umol/L

Exclusion Criteria:

* Have dementia or altered mental status that would prohibit informed consent
* Have previously received treatment for HCV infection (i.e. are currently treatment naïve)
* Have any condition which would deem the patient ineligible for combination therapy with pegylated IFN or ribavirin. This includes pregnancy, significant cardiac, renal or autoimmune disease, severe depression or psychosis, and previous organ transplantation
* Cirrhosis or liver failure as evidenced by clinical (cutaneous stigmata of chronic liver disease, ascites, encephalopathy), ultrasonic (cirrhotic appearance of liver, ascites) or biochemical (platelet count >150 x 109/L, bilirubin <25 umol/L, albumin >35 g/L) evidence, routinely collated in all patients diagnosed with HCV
* Any condition which would preclude the use of rimantadine. This comprises significant renal impairment (creatinine >150), pregnancy, epilepsy or history of unexplained seizures
* Have any other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Chief Investigators, would make the patient inappropriate for this study. This includes the presence of end stage liver disease (cirrhosis), and HIV infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatitis c virus infection who are attending the department of hepatology for treatment with standard combination therpay
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: mark aldersley, mbbs phd, Principal Investigator — national health service; lynsey corless, mbchb phd, Principal Investigator — national health service; stephen griffin, bsc phd, Principal Investigator — University of Leeds
Locations (1):
- St James University Hospital, Leeds, West Yorkshire, United Kingdom